CLINICAL TRIAL: NCT06422533
Title: Ceftolozane/Tazobactam vs. Piperacillin/Tazobactam for the Treatment of Bacteremia Due to Enterobacteriaceae and Pseudomonas Aeruginosa in Hemato-oncological Patients With Severe Neutropenia and Fever: Non-inferiority Study
Brief Title: Ceftolozane/Tazobactam vs. Piperacillin/Tazobactam for the Treatment of Bacteremia in Hemato-oncological Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Patricia Cornejo Juarez, Principal Investigator, Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI0565-2023
Record Dates: First submitted 2024-04-25; First posted 2024-05-21 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Hematologic Neoplasms; Neutropenia
Keywords: ceftolozane/tazobactam; piperacillin/tazobactam; neutropenia; hematologic neoplasms
MeSH Terms: conditions — Hematologic Neoplasms; Neutropenia | interventions — ceftolozane, tazobactam drug combination; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Intervention Model Description: Randomized, open, non-inferiority clinical trial comparing 1:1 two antibiotics, piperacillin/tazobactam vs. ceftolozane/tazobactam
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ceftolozane/tazobactam (Experimental): Ceftozolane/tazobactam (C/T) is a combination antibiotic with a new cephalosporin, structurally similar to ceftazidime, plus tazobactam. The FDA approved This known beta-lactamase inhibitor in 2018 to treat intra-abdominal and complicated urinary infections. In 2019, its indication was expanded to nosocomial pneumonia and those associated with mechanical ventilation. In Mexico, it was approved for marketing in June 2019. C/T has broad-spectrum activity since it has action against ESBL-producing Enterobacteria and MDR P. aeruginosa. Studies carried out in the real world using this antibiotic in patients with hematological malignancies have demonstrated clinical success in reports and case series, considered a therapeutic option in patients with Enterobacteriaceae and P. aeruginosa infections, particularly in MDR pathogens.
  Interventions: Drug: Ceftolozane/tazobactam
- Piperacillin/tazobactam (Active Comparator): At our hospital, Piperacillin/tazobactam is the primary drug used as an empirical treatment in patients with severe neutropenia and fever, according to Clinical Practice Guidelines for the use of antimicrobial agents in neutropenic patients with cancer.
  Interventions: Drug: Piperacillin/tazobactam

INTERVENTIONS:
Drug: Ceftolozane/tazobactam — Ceftolozane/tazobactam 1.5 g tid IV infusion for 1 hour during 5 to 7 days
  Other Names: Zerbaxa
  Arms: Ceftolozane/tazobactam
Drug: Piperacillin/tazobactam — Piperacillin/tazobactam 4.5 g qid IV infusion for 30 minutes during 5 to 7 days
  Other Names: Tazocin; Pipertazo; Tazonam; Tazovak
  Arms: Piperacillin/tazobactam

SUMMARY:
Patients with hematological malignancies receive highly myelotoxic chemotherapy regimens that cause periods of severe myelosuppression, which places them at high risk of developing bacteremia.

At a global level, a very significant increase in multidrug-resistant (MDR) Gram-negative microorganisms, particularly Enterobacteriaceae producing extended-spectrum beta-lactamases (ESBL) and MDR P.aeruginosa, have been described during the last decade. Among the strategies to reduce bacterial resistance, ceftolozane/tazobactam (C/T) as a "carbapenem-sparing" antibiotic has been proposed.

C/T has broad-spectrum activity since it has action against ESBL-producing Enterobacteriaceae and MDR P. aeruginosa. Studies carried out in the real world using this antibiotic in patients with hematological malignancies have demonstrated clinical success in reports and case series, considered a therapeutic option in patients with Enterobacteriaceae and P. aeruginosa infections, particularly in MDR pathogens.

At the National Cancer Institute (in Spanish, Instituto Nacional de Cancerologia), Gram-negative bacilli have been identified for more than 20 years as the pathogens most frequently associated with bacteremia. Escherichia coli occupies the first place in 25% (41% ESBL), followed by Klebsiella spp. in 5.6% (11.2% ESBL) and P. aeruginosa in 5.6% (11.2% MDR). The protocol for approaching and treating hematological malignancy patients with severe neutropenia and fever is to initiate an antimicrobial regimen with piperacillin/tazobactam (P/T). In patients who persist with fever after 48 to 72 hours of starting antibiotics, who present with clinical deterioration, or in whom P/T-resistant bacteria are identified, this is escalated to carbapenem.

Therefore, it is proposed to compare the clinical and microbiological response in patients with hematological malignancies who present with severe neutropenia and fever and who present clinical data of bacteremia, with empirical treatment with C/T vs. P/T, trying to reduce the use of carbapenems in this group of patients.

DETAILED DESCRIPTION:
At a global level, a very significant increase in multidrug-resistant (MDR) Gram-negative microorganisms has been described during the last decade, particularly Enterobacteriaceae producing extended-spectrum beta-lactamases (ESBL) and MDR Pseudomonas aeruginosa. This is directly related to the use of broad-spectrum antimicrobials, particularly carbapenems. Among the strategies to reduce bacterial resistance, using ceftolozane/tazobactam (C/T) as a "carbapenem-sparing" antibiotic is proposed. C/T has been administered in hemato-oncological patients with severe neutropenia, colonized by resistant strains in centers with a high prevalence of Enterobacteriaceae-ESBL and P. aeruginosa MDR.

The study's purpose is to demonstrate non-inferiority between ceftolozane/tazobactam vs. piperacillin/tazobactam for patients with hematological malignancies who present severe neutropenia and fever, including those patients who have bacteremia due to Enterobacteriaceae and Pseudomonas aeruginosa. C/T is a combination antibiotic with a new cephalosporin, structurally similar to ceftazidime, plus tazobactam. The FDA approved This known beta-lactamase inhibitor in 2018 to treat intra-abdominal and complicated urinary infections. In 2019, its indication was expanded to nosocomial pneumonia and those associated with mechanical ventilation. In Mexico, it was approved for marketing in June 2019. C/T has broad-spectrum activity since it has action against ESBL-producing Enterobacteria and MDR P. aeruginosa. Studies carried out in the real world using this antibiotic in patients with hematological malignancies have demonstrated clinical success in reports and case series, considered a therapeutic option in patients with Enterobacteriaceae and P. aeruginosa infections, particularly in MDR pathogens.

At the National Cancer Institute, Gram-negative bacilli have been identified for more than 20 years as the pathogens most frequently associated with bacteremia, with Escherichia coli occupying first place at 25% (41% ESBL), followed by Klebsiella sp. in 5.6% (11.2% ESBL), and P. aeruginosa in 5.6% (11.2% MDR). The protocol for approaching and treating hemato-oncological patients with severe neutropenia and fever is to initiate an antimicrobial regimen with piperacillin/tazobactam (P/T) if they are hemodynamically stable. In patients who persist with fever after 48 to 72 hours of starting antibiotics, who present with clinical deterioration, or in whom P/T-resistant bacteria are identified, this is escalated to a carbapenem (usually meropenem).

A randomized, open, non-inferiority clinical trial comparing 1:1 two antibiotics, P/T vs. C/T, for the treatment of severe neutropenia and fever and/or developing Enterobacteriaceae or P. aeruginosa bacteremia in patients with hematologic malignancies

Methodological strategies All patients who come to the National Cancer Institute with signs of severe neutropenia (polymorphonuclear cells <500 cells/mm3) and fever (≥38.3 degrees Celsius in one measure or ≥38 degrees Celsius in at least two measures) will be considered for inclusion. Blood cultures will be taken upon admission (catheter and peripheral in those with the same), or two peripherals with a difference of 15 minutes between each one. Blood cultures will be requested before signing the informed consent since they are part of the initial approach to these patients, regardless of whether they enter the study. They will be taken before the administration of antimicrobials.

Medical staff from the infectious disease department will evaluate the inclusion and exclusion criteria and invite the candidate to the study.

If the patient accepts, they will be provided informed consent to review it in detail, explaining any doubts. If they agree to participate, the corresponding signatures will be made.

Randomization will be done based on a stratified method in two groups: Group 1, patients with leukemia, and Group 2, patients with other hemato-oncological pathologies. They will be randomized into ten blocks and divided into the two groups above.

The administration of the P/T or C/T antimicrobial regimen will begin depending on the group to which they have been assigned, following the manufacturer's instructions and according to the administration standards at INCan.

The clinical and microbiological response will be evaluated in the first 72-96 hours (taking randomization as day +1), defined as patient survival plus resolution of fever plus sterilization of blood cultures (taken within the first 72-96 hours).

If patients have been fever-free for at least 48 hours and have no growth in blood cultures, they will receive at least five days of antibiotic treatment.

The administration time will be at least seven days in patients with P. aeruginosa or Enterobacteriaceae growth in blood cultures.

Patients whose blood cultures report growth of bacteria different from the previous ones, yeast, or polymicrobial growth will be excluded from the study.

Treatment failure will be considered, and the following will be included in the intention-to-treat analysis:

* If the growth in the blood culture is Enterobacteriaceae or P. aeruginosa, resistant to the antibiotic assigned.
* There is growth of the same bacteria in control blood cultures taken 72-96 hours after starting antibiotics.
* If, during treatment, the patient presents signs of hemodynamic instability, respiratory failure, clinical deterioration, or septic shock, changing the antimicrobial regimen will be considered.

The following will be considered a relapse and will be included in the intention-to-treat analysis:

* When the same microorganism is isolated at the beginning, it grows in blood cultures after having negative blood cultures.
* Or in the first 30 days after completing the antibiotic regimen, considering the resolution of the primary infectious focus.

During treatment, they will not be able to receive any other Gram-negative antibiotic except prophylaxis against P. jirovecii (400/80 mg/day TMP/SMX or 800/160 mg every 48 h).

The number of days of antibiotics will be counted. It will be documented when an antibiotic is modified and the reason for the change (microbiological failure, clinical deterioration, drug-related adverse events, and others). The appearance of diarrhea will be monitored, and Glutamate dehydrogenase (GDH) and toxin for Clostridiodes difficile will be requested.

Patients will be evaluated daily until fever resolution and until hospital discharge (if this occurs in the first 14 days), recording fever and adverse events, including diarrhea, leukocytes, and neutrophils. Follow-up will be carried out until day +30 from the patient's inclusion in the study. If the patient is discharged before this date, a telephone call will be made on day +30 to verify the clinical status.

The evolution will be classified as alive without infection, alive with clinical or microbiological data of infection, also considering C. difficile infection, dead from infection without neutropenia, dead from infection with neutropenia, dead from terminal illness, or dead from another cause.

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years old
* Diagnosis of any hematological malignancy
* Severe neutropenia (polymorphonuclear <500 cells/mm3)
* Fever (≥38.3 degrees Celsius in one measure, or ≥38 degrees Celsius in at least two measures)
* Median arterial pressure ≥65 mmHg on admission
* A life expectancy ≥ 5 days
* Agree to participate in the study

Exclusion Criteria:

* Known hypersensitivity to cephalosporins or anaphylaxis with beta-lactams
* Clinical signs related to hemodynamic instability
* Concomitant use of another antibiotic with activity against Gram-negatives (except Trimethoprim/Sulfamethoxazole (TMP/SMX) as prophylaxis for P. jirovecii
* Patients with end-stage chronic renal failure (<10 ml/min by creatinine clearance-ACCr) or on renal replacement therapy.
* Patients with grade IV mucositis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Mortality of all patients at day 30 | Day 30
  To assess the number of patients who will be alive or dead in the first 30 days. On day 30, a physical visit will be made to the patient's bedside if the patient is hospitalized. If the patient is not hospitalized, the clinical record will be evaluated, and one of the investigators will make a phone call to ensure the patient's status for that date.

SECONDARY OUTCOMES:
Microbiological response through the sterilization of repeated blood cultures take | Day 3 to day 4
  Number of patients that will have repeated blood cultures sterilized (no growth of the same bacteria isolated in the first set of blood cultures taken in day 1).
Clinical response measured through fever resolution | Day 4
  The presence of fever (>38 Celsius degree) will be evaluated according to nursing records that are carried out three times a day (morning, afternoon, and night shifts). Clinical failure will be considered when the patient persists with fever (>38 Celsius degrees) on day four after starting the antimicrobial regimen. Clinical success will be considered when the fever resolves between day 1 and day 3 of starting antibiotics.

OTHER OUTCOMES:
Clostridioides difficile infection documented through toxin/GDH C. difficile test in those patients who develop diarrhea, abdominal pain and/or distended abdomen. | Day 1 to day 30
  Number of patients who develop diarrhea or abdominal pain or distended abdomen, with a test positive for C. difficile (toxin/GDH C. difficile test).

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Cornejo-Juarez, M.D.,M.Sc., Principal Investigator — Instituto Nacional de Cancerología, Mexico
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) could be shared with other researchers.
Supporting Information: Study Protocol, ICF
Time Frame: The data will become available at the end of the study. The plan is to finish the analysis and write the manuscript at the end of 2025.
Access Criteria: The data requisition must be carried out with a solid foundation for which the information will be used. The investigators and sub-investigators will review the criteria.

REFERENCES:
- [Background] Karaiskos I, Giamarellou H. Carbapenem-Sparing Strategies for ESBL Producers: When and How. Antibiotics (Basel). 2020 Feb 5;9(2):61. doi: 10.3390/antibiotics9020061. PMID 32033322
- [Background] Xie O, Cisera K, Taylor L, Hughes C, Rogers B. Clinical syndromes and treatment location predict utility of carbapenem sparing therapies in ceftriaxone-non-susceptible Escherichia coli bloodstream infection. Ann Clin Microbiol Antimicrob. 2020 Nov 30;19(1):57. doi: 10.1186/s12941-020-00400-z. PMID 33256752
- [Background] Giacobbe DR, Bassetti M, De Rosa FG, Del Bono V, Grossi PA, Menichetti F, Pea F, Rossolini GM, Tumbarello M, Viale P, Viscoli C; ISGRI-SITA (Italian Study Group on Resistant Infections of the Societa Italiana Terapia Antinfettiva). Ceftolozane/tazobactam: place in therapy. Expert Rev Anti Infect Ther. 2018 Apr;16(4):307-320. doi: 10.1080/14787210.2018.1447381. Epub 2018 Mar 9. PMID 29493397
- [Background] Shortridge D, Pfaller MA, Castanheira M, Flamm RK. Antimicrobial Activity of Ceftolozane-Tazobactam Tested Against Enterobacteriaceae and Pseudomonas aeruginosa with Various Resistance Patterns Isolated in U.S. Hospitals (2013-2016) as Part of the Surveillance Program: Program to Assess Ceftolozane-Tazobactam Susceptibility. Microb Drug Resist. 2018 Jun;24(5):563-577. doi: 10.1089/mdr.2017.0266. Epub 2017 Oct 17. PMID 29039729
- [Background] Pfaller MA, Bassetti M, Duncan LR, Castanheira M. Ceftolozane/tazobactam activity against drug-resistant Enterobacteriaceae and Pseudomonas aeruginosa causing urinary tract and intraabdominal infections in Europe: report from an antimicrobial surveillance programme (2012-15). J Antimicrob Chemother. 2017 May 1;72(5):1386-1395. doi: 10.1093/jac/dkx009. PMID 28165526
- [Background] Livermore DM, Mushtaq S, Meunier D, Hopkins KL, Hill R, Adkin R, Chaudhry A, Pike R, Staves P, Woodford N; BSAC Resistance Surveillance Standing Committee. Activity of ceftolozane/tazobactam against surveillance and 'problem' Enterobacteriaceae, Pseudomonas aeruginosa and non-fermenters from the British Isles. J Antimicrob Chemother. 2017 Aug 1;72(8):2278-2289. doi: 10.1093/jac/dkx136. PMID 28520867
- [Background] Pfaller MA, Shortridge D, Sader HS, Flamm RK, Castanheira M. Ceftolozane-tazobactam activity against drug-resistant Enterobacteriaceae and Pseudomonas aeruginosa causing healthcare-associated infections in Australia and New Zealand: Report from an Antimicrobial Surveillance Program (2013-2015). J Glob Antimicrob Resist. 2017 Sep;10:186-194. doi: 10.1016/j.jgar.2017.05.025. Epub 2017 Jul 19. PMID 28735046
- [Background] Pfaller MA, Shortridge D, Sader HS, Gales A, Castanheira M, Flamm RK. Ceftolozane-tazobactam activity against drug-resistant Enterobacteriaceae and Pseudomonas aeruginosa causing healthcare-associated infections in Latin America: report from an antimicrobial surveillance program (2013-2015). Braz J Infect Dis. 2017 Nov-Dec;21(6):627-637. doi: 10.1016/j.bjid.2017.06.008. Epub 2017 Sep 21. PMID 28941394
- [Background] Seifert H, Korber-Irrgang B, Kresken M; German Ceftolozane/Tazobactam Study Group. In-vitro activity of ceftolozane/tazobactam against Pseudomonas aeruginosa and Enterobacteriaceae isolates recovered from hospitalized patients in Germany. Int J Antimicrob Agents. 2018 Feb;51(2):227-234. doi: 10.1016/j.ijantimicag.2017.06.024. Epub 2017 Jul 10. PMID 28705666
- [Background] Fernandez-Cruz A, Alba N, Semiglia-Chong MA, Padilla B, Rodriguez-Macias G, Kwon M, Cercenado E, Chamorro-de-Vega E, Machado M, Perez-Lago L, Garcia de Viedma D, Diez Martin JL, Munoz P. A Case-Control Study of Real-Life Experience with Ceftolozane-Tazobactam in Patients with Hematologic Malignancy and Pseudomonas aeruginosa Infection. Antimicrob Agents Chemother. 2019 Jan 29;63(2):e02340-18. doi: 10.1128/AAC.02340-18. Print 2019 Feb. PMID 30530598
- [Background] Bergas A, Albasanz-Puig A, Fernandez-Cruz A, Machado M, Novo A, van Duin D, Garcia-Vidal C, Hakki M, Ruiz-Camps I, Del Pozo JL, Oltolini C, DeVoe C, Drgona L, Gasch O, Mikulska M, Martin-Davila P, Peghin M, Vazquez L, Laporte-Amargos J, Dura-Miralles X, Pallares N, Gonzalez-Barca E, Alvarez-Uria A, Puerta-Alcalde P, Aguilar-Company J, Carmona-Torre F, Clerici TD, Doernberg SB, Petrikova L, Capilla S, Magnasco L, Fortun J, Castaldo N, Carratala J, Gudiol C. Real-Life Use of Ceftolozane/Tazobactam for the Treatment of Bloodstream Infection Due to Pseudomonas aeruginosa in Neutropenic Hematologic Patients: a Matched Control Study (ZENITH Study). Microbiol Spectr. 2022 Jun 29;10(3):e0229221. doi: 10.1128/spectrum.02292-21. Epub 2022 Apr 27. PMID 35475683
- [Background] Criscuolo M, Trecarichi EM. Ceftazidime/Avibactam and Ceftolozane/Tazobactam for Multidrug-Resistant Gram Negatives in Patients with Hematological Malignancies: Current Experiences. Antibiotics (Basel). 2020 Feb 3;9(2):58. doi: 10.3390/antibiotics9020058. PMID 32028615
- [Background] Marchesi F, Toma L, Di Domenico EG, Cavallo I, Spadea A, Prignano G, Pimpinelli F, Papa E, Terrenato I, Ensoli F, Mengarelli A. Ceftolozane-Tazobactam for Febrile Neutropenia Treatment in Hematologic Malignancy Patients Colonized by Multi-Resistant Enterobacteriaceae: Preliminary Results from a Prospective Cohort Study. Mediterr J Hematol Infect Dis. 2020 Sep 1;12(1):e2020065. doi: 10.4084/MJHID.2020.065. eCollection 2020. No abstract available. PMID 32952976
- [Background] Clerici D, Oltolini C, Greco R, Ripa M, Giglio F, Mastaglio S, Lorentino F, Pavesi F, Farina F, Liberatore C, Castiglion B, Tassan Din C, Bernardi M, Corti C, Peccatori J, Scarpellini P, Ciceri F, Castagna A. The place of ceftazidime/avibactam and ceftolozane/tazobactam for therapy of haematological patients with febrile neutropenia. Int J Antimicrob Agents. 2021 Jun;57(6):106335. doi: 10.1016/j.ijantimicag.2021.106335. Epub 2021 Apr 7. PMID 33838223